CLINICAL TRIAL: NCT05564897
Title: Phase II Single Center Open-Label Single-Arm Study of the Safety and Efficacy of Oncolytic Adenovirus H101 Combined With PD-1 Inhibitor in Patients With Non-muscle-invasive Bladder Cancer Who Failed BCG Therapy
Brief Title: Oncolytic Adenovirus Combined With PD-1 Inhibitor in Patients With Non-muscle-invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Hua, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUCAS-030
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer, oncolytic adenovirus, intravesical therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of H101 with Camrelizumab treatment (Experimental): Patients receive a combination therapy of PD-1 inhibitor Camrelizumab with oncolytic adenovirus H101 for up to 1 years. Camrelizumab are administered at dose of 200 mg i.v. every 3 weeks. H101 are instilled intravesically with a dose of 5×10*11 Vp in a 50 mL normal saline solution via a catheter, and dwell time is 1 to 2 hours,. Intravesical H101 is instilled weekly for 6 weeks for both induction and maintenance treatments.
  Interventions: Drug: H101, Camrelizumab

INTERVENTIONS:
Drug: H101, Camrelizumab — Patients receive a combination therapy of Camrelizumab 200 mg i.v. every 3 weeks with intravesical H101 with a dose of 5×10*11 Vp weekly for 6 weeks for both induction and maintenance treatments up to 1 years.

SUMMARY:
H101 is an E1B55KD deleted oncolytic adenovirus, which is the first and only adenovirus to be approved by China State Food and Drug Administration in 2005 for treating head and neck cancer. The objective of this phase II clinical trial is to investigate the safety and efficacy of H101 combined with PD-1 inhibitor Camrelizumab in patients with non-muscle-invasive bladder cancer who failed BCG therapy.

DETAILED DESCRIPTION:
CHUCAS-030 (Cancer Hospital, University of Chinese Academy of Sciences) is a phase II trial conducted at Cancer Hospital, University of Chinese Academy of Sciences in the Zhejiang Province, China. Eligible patients are 18 to 80 years old with non-muscle-invasive bladder cancer who has previously failed BCG therapy and refuse cystectomy. Patients receive a combination therapy of PD-1 inhibitor Camrelizumab with oncolytic adenovirus H101 for up to 1 year. Camrelizumab are administered at dose of 200 mg i.v. every 3 weeks. H101 are instilled intravesically after 14 days from the most recent biopsy and in the absence of any evidence of hematuria with a fixed dose of 5×10*11 Vp in a 50 mL normal saline solution via a catheter, and dwell time is 1 to 2 hours, and patients are encouraged to reposition to maximize bladder surface exposure. Intravesical H101 is instilled weekly for 6 weeks for both induction and maintenance treatments. Patients who experienced unacceptable toxicities or clinical or documented progressive disease are discontinued from the study. The duration of any objective response is measured from the date the initial response is observed to the date that disease progression is observed. Response assessment with cystoscopy, bladder biopsy of visually positive lesions and urine cytology are first evaluated after induction at 3 months. Patients with complete response (CR) at 3 months receive no intervention and are reevaluated at 6 months. Patients with stable disease (SD) receive maintenance treatment at 3 to 4 months. Patients with progressive disease (PD) are deemed non-responders and strongly counseled to reconsider cystectomy or alternative treatment. Patients with CR at 6 months receive maintenance treatment (weekly treatments for 6 weeks). All patients were followed up until death from any cause.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 ~80 years old.
2. Patients who are diagnosed pathologically with urothelial carcinoma of non-muscle invasive bladder cancer and have previously failed BCG therapy and refused cystectomy.
3. Performance status: Eastern Cooperative Oncology Group performance 0-2.
4. Life expectancy more than 3 months.
5. Patients have adequate organ function, accord with following criteria: A. blood routine: Hemoglobin≥90g/L, absolute neutrophil count≥1.5×10*9/L, platelet count ≥ 80×109/L; B. Biochemical tests: total bilirubin is less than 1.5 times upper limit of normal, alanine aminotransferase and aspartate aminotransferase are less than 2.5 times upper limit of normal; C. creatinine less than 1.25 times upper limit of normal.
6. Patients agree to use adequate contraception in the period of trial and need negative pregnancy test in childbearing potential women.
7. Participant sign an institutional review board-approved, protocol specific informed consent form in accordance with institutional guidelines.

Exclusion Criteria:

1. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
2. Organs failure.
3. ECOG >2.
4. Serious/active infection.
5. Autoimmune disorders or immunodeficiency diseases.
6. Patients with allergic constitution, or other disease need take drugs of immunosuppressant or corticosteroids.
7. Uncontrolled hypertension.
8. Myocardial ischemia (more than grade II ) or myocardial infarction or uncontrolled arrhythmia.
9. Cardiac insufficiency of grade III to IV according to NYHA criteria, or left ventricular ejection fraction (LVEF) <50%.
10. Coagulation disorders, tendency of haemorrhage, undergoing thrombolytic or anticoagulant therapy.
11. Unhealed wounds, or fractures.
12. With a history of psychotropic drug abuse or mental disorders.
13. Prior systemic therapies with any antitumor agents within 4 weeks.
14. With other uncurable cancers simultaneously.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) | One year
  CR is deemed by negative cystoscopy, urine cytology, and bladder biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, Ph.D.；M.D., Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Hua Wang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No